CLINICAL TRIAL: NCT01459692
Title: Reduction and Prevention of Seizure Occurrence From Exposure to Auditory Stimulation in Individuals With Neurological Handicaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: MIND Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR15863
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Seizures; Epilepsy
Keywords: Seizures; Epilepsy; Auditory Stimulation; Music
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group - No Music Exposure (No Intervention): Subjects that were assigned to the control group of the study were not exposed to music.
- Music Exposure (Experimental): The treatment subjects were randomly assigned to receive nightly exposure to music at periodic intervals between the hours of 9:00 PM and 8:00 AM.
  Interventions: Other: Music Exposure

INTERVENTIONS:
Other: Music Exposure — Twenty-seven subjects were randomly assigned to receive nightly exposure to music at periodic intervals between the hours of 9:00 PM and 8:00 AM.
  Arms: Music Exposure

SUMMARY:
Neurologically-impaired individuals may have significant neurologic morbidity related to epilepsy and seizure disorders. Finding safe, noninvasive methods of decreasing seizures, and potentially reversing the epileptogenic process, is of paramount importance in improving the lives of those with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Thad E. Saleeby Center
* Epilepsy or seizure disorder
* At least one year of detailed seizure reporting prior to study starting date

Exclusion Criteria:

* Severe hearing impairment

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Changes in seizure rates | 3 years
  Main Outcome Measure: The effect of exposure to the auditory stimulus on seizure frequency. Changes in seizure rates from baseline to treatment years were determined and statistically compared within the treatment and control groups, as well as between the groups to assess efficacy of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Turner, MD, MSCR, Principal Investigator — Medical University of South Carolina; Mark Bodner, Ph.D., Principal Investigator — MIND Research Institute
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Bodner M, Turner RP, Schwacke J, Bowers C, Norment C. Reduction of seizure occurrence from exposure to auditory stimulation in individuals with neurological handicaps: a randomized controlled trial. PLoS One. 2012;7(10):e45303. doi: 10.1371/journal.pone.0045303. Epub 2012 Oct 11. PMID 23071510